CLINICAL TRIAL: NCT04605354
Title: Epidemiological and Clinical Description of Women Living With HIV in Selected Countries of Latin America
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Helios Salud (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: Women living with HIV in LATAM
Record Dates: First submitted 2020-09-08; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: HIV-1-infection; Hiv
Keywords: Women; Latin America
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study that uses ecological data from (1) PLWHIV under care at 31st December 2017, and (2) from yearly admissions to care occurred during 2013 - 2017, from centers belonging to LAW-HIV.

DETAILED DESCRIPTION:
General Aims Aim 1: Epidemiological and clinical description of women that receive HIV care in selected countries of Latin America.

Aim 2: Management of HIV infection during pregnancy in women from selected countries of Latin America.

Countries: Argentina, Bolivia, Chile, Colombia, Costa Rica,Ecuador, Guatemala, Honduras, México, Peru, Dominican, Republic, Uruguay, and Venezuela.

Background & Relevance of this specific study:

Research Approach:

The Latin American Workshop for HIV Studies (LAW-HIV) includes more than 70 clinical centers belonging to 14 Spanish speaking countries from the region. It gathers aggregate information form more than 116.000 people living with HIV under care, from which 25,802 are women.

These numbers represent roughly a fifth of the total estimated female under care in these countries.

Specific aims from overall aim 1:

The investigators will determine at center, national and regional level:

* The age distribution of women under care for HIV infection as of December 31st, 2017.
* The fraction of women under care who are receiving ART as of December 31st, 2017.
* The age distribution of women admitted to care for years 2013, 2014, 2015, 2016 and 2017.
* The fraction of admitted women that start ART during the first year after admission, by year of admission.
* Frequency of selected type of drugs (for backbone and 3rd drug) used for the first cART, by year of admission and age group.
* The frequency late and very late presenters (CD4) in women admitted according to year of admission and age group.
* The fraction of women alive, retained to care, retained to ART, and with virologic suppression at one year of follow up, from admissions occurred in 2016.

Specific aims from overall aim 2:

The investigators will determine:

* The fraction of women with HIV diagnosis occurred as consequence of the pregnancy.
* Earliest CD4 level and viral load in pregnant women under care by HIV.
* The fraction of women that suspend ART during pregnancy; frequency of each scheme of ART used previous the conception; and change of scheme (3rd drug and backbone).
* The fraction of women whose pregnancy ended in term, preterm or as abortion.
* The fraction of women retained in control post pregnancy.
* The fraction of women that suspended breastfeeding Data Collection & Quality:

Study Design:

A cross-sectional study that uses ecological data from (1) People living with HIV under care at 31st December 2017, and (2) from yearly admissions to care occurred during 2013 - 2017, from centers belonging to LAW-HIV. Data will be weighted by the expected population under care in each country considering attributes of the centers (private/public). Weighted outcomes at strata level from each center will be meta-analyzed considering three levels of heterogeneity (stratum, center, and country) and modeled through multilevel regression models to allow adjustment for covariables of the stratum. In the case of admissions to care, a time series analysis will be implemented.

Data collection and quality control:

Data collection will be carried out through a spreadsheet sent to centers that agree to participate. Two different spreadsheets will be sent, one for each general aim of the study (see the annex at the complete project). A quality check will be implemented at three stages: (1) at the moment of receiving each spreadsheet back; (2) previous to analysis, where the consistency of information across strata from different sections will be assessed; and (3) identifying outlier values from outcomes at the centers level, using expert criteria.

Data information included:

1. Center description (health care staff, ART & labs (e.g. viral load determinations) availability)
2. Demographic and clinical features of women under control and admitted (age, CD4, the scheme of ART, retention to care, retention to ART, virologic suppression one year later the admission).
3. Clinical features of pregnant women under care infected by HIV.

Total duration: 18 months.

ELIGIBILITY:
* All Latin American HIV care centers from any Spanish speaking country are invited to participate in the LAW-HIV.
* Only centers that provide a minimum of information (at least sections 1 and 2 from the datasheet for aim 1) will be included in the analysis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the overall aim 1, the investigators expected to include information about 25,816 women under care, and between 6,000 and 7,500 women admitted during 2013 - 2017 (depending on the sub-analysis), from 14 countries and 79 centers.
  For the overall aim 2, the investigators expect to include aggregated information from roughly 400 pregnant females, from at least ten countries. It is worth noticing that the analytic unit corresponds to the information at the stratum level and depending on the disposition of the information in the database, the total numbers of strata will vary between approximately 400 to 8.000.
Sampling Method: Non-Probability Sample
Enrollment: 25816 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiological and clinical description of women that receive HIV care in selected countries of Latin America. | 1 year
  1.1. In women admitted to care between years 2013-2017, the trend in the:
  * distribution of ages;
  * proportion of late presenters (CD4).
  * proportion that start ART during the first year after admission;
  * schemes of ART used for the first ART.
  1.2. Proportion of women alive, retained to care, retained to ART, and with virologic suppression at one year of follow up, from admissions occurred in 2016.
Management of HIV infection during pregnancy in women from selected countries of Latin America. | 1 year
  2. In women that finished their pregnancy at any moment during 2019:
  * Proportion with HIV diagnosis as consequence of the pregnancy.
  * Earliest CD4 level.
  * Proportion that suspended ART during pregnancy
  * Frequency of each scheme of ART used previous the conception
  * Change of scheme of ART
  * Proportion whose pregnancy ended in term
  * Proportion retained in care during the first 6 months after pregnancy
  * Proportion that suspended breastfeeding during the first 3 months after pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Cassetti, MD, Principal Investigator — Helios Salud
Locations (1):
- Helios Salud, Buenos Aires, Argentina